CLINICAL TRIAL: NCT02347241
Title: Infant Special Program for In Hospital Resuscitation Education in the Delivery Room - INSPIRE-D
Brief Title: Infant Special Program for In Hospital Resuscitation Education in the Delivery Room
Acronym: INSPIRE-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Theresa Mariero Olasveengen, Researcher, Oslo University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013/12769
Record Dates: First submitted 2015-01-12; First posted 2015-01-27 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Hypoxia, in Liveborn Infant; Neonatal Asphyxia; Neonatal Bradycardia
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control period (No Intervention): Assessment of resuscitation quality and clinical outcomes prior to educational intervention
- Educational intervention (Experimental): Assessment of resuscitation quality and clinical outcomes after educational intervention consisting of debriefing and rolling refreshers.
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — Educational Debriefings and High frequency training and team reflection
  Arms: Educational intervention

SUMMARY:
The overall objective is to determine whether a bundled In-hospital Newborn Resuscitation Edu-cation intervention (INSPIRE-D) improves process of care associated with improved newborn survival and neurologic outcomes.

DETAILED DESCRIPTION:
This prospective interventional trial will be conducted in the delivery unit at OUS. The planned studies consist of five distinct phases with step-wise interventions; 1) baseline data collection, 2) introducing educational debriefing, 3) intensive run-in/rolling-refresher phase, 4) INSPIRE-D phase and lastly 5) evaluation phase.

Phase 1: The baseline data collection phase

1. Needs assessment/questionnaires from participating healthcare providers will be collected which include demographic data such as sex, age, education, and work experience, as well as exposure to resuscitation training, simulation, self-perceived confidence and suggestions for further training/educational topics.
2. Observations of the newborn in the resuscitation bays will be done by video recordings and supplemented by resuscitation records, hospital quality improvement data and medical records. Data points to be collected of the newborn are demographics, gestational age, physiological parameters such as heart rate and respirations/oxygenation, Apgar score, interventions performed, and outcomes during and at discharge from hospital.
3. The healthcare providers adherence to guidelines in neonatal resuscitation (both technical and non-technical skills like team collaboration) will be evaluated by examining the video recordings and scored by validated scoring systems formerly tested with good intra- and inter-rater reliability. The scoring systems is adapted to guidelines from the Norwegian Council of Resuscitation and retested for intra- and inter-rater reliability.

Phase 2: Intervention Phase with Educational Debriefings

1. Educational debriefings of healthcare providers involved in clinical situations with newborn resuscitation: Selected resuscitation events will be debriefed facilitated by a study team member with special competence in facilitation and an instructor in neonatal resuscitation. The debriefing will be held depending on clinical schedule and availability, to discuss process of care, performance, and provide education to multidisciplinary staff with advocacy/inquiry debriefing techniques.
2. For healthcare providers; cont¬inued needs assessment and prospective observations by video-recordings in resuscitation bays to document quality of care.
3. Baseline skills assessment will be collected using a novel manikin, the Newborn Lung Simulator. Healthcare providers will be presented for a mini-simulation with a compromised newborn and asked to perform high quality resuscitation. The performance and adherence to guidelines will be evaluated and retested after the intervention.

Phase 3 - Intensive run-in of high frequency training and team reflection: "The rolling refresher phase"

1. In this phase training triggers are identified at the start of each day shift. A careful consideration of perinatal factors of both mother and infant will identify "high risk" deliveries with babies who may need resuscitation. If no risk deliveries are identified, a random Healthcare Provider team among the present staff will be selected.
2. "Just-in-time" and "just-in-place" training; the novel "Rolling refresher", will be introduced (target >80% of staff) at the beginning of day shifts. Health Care Providers caring for labouring mothers with training triggers will be identified and exposed to "low dose" simulation-based "just-in-time" and "just-in-place" skills training. The short training session (<10 minutes) will take place on-site in the resuscitation bay with relevant topics such as; timely assessment of need for intervention, effective assisted ventilations on a Newborn Lung Simulator. We will use observations from the video-films to target training with focus on rapid evaluation of respiratory distress, correct ventilation technique and use of pulse oximetry.
3. Continued simulation training will be based on problem areas identified from baseline. Performance during simulation training will be evaluated and registered.
4. Educational debriefings will continue, as in Phase 2
5. Continued needs assessment and prospective observations in resuscitation bays to document provider confidence, simulation performance and quality of care during implementation of the INSPIRE-D bundle described above.

Phase 4: Continued INSPIRE-D bundle. After successful implementation defined as >80% of staff having been through at least one "just-in-time and just in place" training session, all interventions above (phase 2 and 3) will continue on routine basis. Continued needs assessment of confidence and performance are repeated as described above.

Phase 5: Evaluation. Evaluation of the INSPIRE-D bundle to identify and define key factors and processes that we prove necessary to ensure timely and effective neonatal resuscitation associated with improved newly born survival and neurologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Neonates that require stabilisation and/or resuscitation such as ventilatory support, medications and/or chest compressions.

Exclusion Criteria:

* Parent or health care provider reserved against study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Quality of neonatal resuscitation (Validated performance score assessed by video analysis) | 12 months
  Validated performance score assessed by video analysis

SECONDARY OUTCOMES:
Clinical outcome - Time to effective respiration | 12 months
Clinical outcome - Time to heart rate > 100 | 12 months
Clinical outcome - Admission to intensive care | 12 months
Health care providers adherence to guidelines and behaviour markers - Self-reported score | 12 months
Health care providers adherence to guidelines and behaviour markers - Simulation score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Theresa M Olasveengen, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Niles DE, Skare C, Foglia EE, Insley E, Cines C, Olasveengen T, Ballester LS, Ades A, Posencheg M, Nadkarni VM, Kramer-Johansen J. Effect of a positive pressure ventilation-refresher program on ventilation skill performance during simulated newborn resuscitation. Resusc Plus. 2021 Feb 16;5:100091. doi: 10.1016/j.resplu.2021.100091. eCollection 2021 Mar. PMID 34223356
- [Derived] Skare C, Boldingh AM, Kramer-Johansen J, Calisch TE, Nakstad B, Nadkarni V, Olasveengen TM, Niles DE. Video performance-debriefings and ventilation-refreshers improve quality of neonatal resuscitation. Resuscitation. 2018 Nov;132:140-146. doi: 10.1016/j.resuscitation.2018.07.013. Epub 2018 Jul 18. PMID 30009926
- [Derived] Skare C, Boldingh AM, Nakstad B, Calisch TE, Niles DE, Nadkarni VM, Kramer-Johansen J, Olasveengen TM. Ventilation fraction during the first 30s of neonatal resuscitation. Resuscitation. 2016 Oct;107:25-30. doi: 10.1016/j.resuscitation.2016.07.231. Epub 2016 Aug 2. PMID 27496260